CLINICAL TRIAL: NCT05190107
Title: Prevalence of Depression, Anxiety and Stress in High School Students: A Survey Study in Western Mexico
Brief Title: Depression, Anxiety and Stress in High School
Status: Completed | Type: Observational
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, GONZALEZ-OJEDA ALEJANDRO, Principal Investigator D, Instituto Mexicano del Seguro Social
Other Study IDs: DASSH
Record Dates: First submitted 2021-12-10; First posted 2022-01-13 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2021-12

CONDITIONS: Depression; Anxiety; Stress
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: DASS-21 scale — Each construct consists of 7 questions. The participants must select the answer that better represents their feelings over the last week in each scenario. Each question has a Likert scale of 4 options where 0 represents "did not apply to me" to 3 "applied to me very much.

SUMMARY:
Background: Social isolation secondary to the pandemic can predispose the population to mental health issues in the future, especially teenagers. The Depression, Anxiety, and Stress Scale (DASS) is a valuable self-report scale since it may be used to screen for anxiety, depression, and stress in one questionnaire. In the last years, it has been observed effective in detecting these symptoms in teenagers.

Aims: Identify the prevalence of depression, anxiety, and stress in high school students during the COVID-19 pandemic This is an observational cross-sectional study.

For this study, the validated Spanish version of DASS-21 will be used. Qualitative variables will be evaluated through central tendencies, such as mean, standard deviation, and frequencies. The inferential analysis of categorical variables will be performed using the chi-squared test, analysis of variance (ANOVA), or Kruskal Wallis test as appropriate. For quantitative variables, Student's t-test or Mann Whitney U test will be performed depending on their distribution.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents from 14 to 22 years old.
* That they voluntarily agree to participate, and consent.

Exclusion Criteria:

* Adolescents with depression, anxiety, and stress disorders previously detected
* Patients in psychiatric treatment for depression, anxiety, or stress.
* Participants who don´t consent to participate

Ages: 14 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Adolescents from 14 to 22 years old with an average age of 16 years are high school students.
Sampling Method: Non-Probability Sample
Enrollment: 3112 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-12-10 (Actual)

PRIMARY OUTCOMES:
Depression Score | Baseline
  the Depression, Anxiety and Stress Scale 21 (DASS-21) is an inventory that will be used to identify the presence and intensity of depressive, anxiety and stress. For depression the cutoff scores are: Normal: 0-9, Mild: 10-12, Moderate:13-20, Severe: 21-27, and Extremely severe: 28-42.
Anxiety Score | Baseline
  the Depression, Anxiety and Stress Scale 21 (DASS-21) is an inventory that will be used to identify the presence and intensity of depressive, anxiety and stress. For anxiety the cutoff scores are: Normal: 0-6, Mild: 7-9, Moderate: 10-14, Severe:15-19, and Extremely severe: 20-42.
Stress Score | Baseline
  the Depression, Anxiety and Stress Scale 21 (DASS-21) is an inventory that will be used to identify the presence and intensity of depressive, anxiety and stress. For stress the cutoff scores are: Normal: 0-10, Mild:11-18, Moderate:19-26, Severe: 27-34, and Extremely severe: 35-42.

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Médico Nacional de Occidente, Guadalajara, Jalisco, Mexico